CLINICAL TRIAL: NCT02819206
Title: Microbiological Diagnosis of Infectious Uveitis to Pathogenic Fastidious Germs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-41; 2012-A01563-40 (Other: ANSM)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uveitis (Other): Patient with a prescription of a microbiologic diagnostic of uveitis
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Detection of bacteria will be performed on a blood sample

SUMMARY:
Our research project is to use a new microbiological diagnostic strategy of uveitis, allowing detection of the fastidious pathogens of infectious Uveitis who are not diagnosed by laboratory methods used in diagnostic routine. This new diagnostic strategy is to automatically detect the presence of a pathogen fastidious in cell culture using the same patient's serum to reveal a positive culture, based on the assumption that this serum contains antibodies specific pathogen tedious.

Finally, the main purpose of this study is to improve the etiological diagnosis of Uveitis by establishing a new diagnostic strategy.

DETAILED DESCRIPTION:
The Mediterranean Infection microbiology laboratory is the national Reference Laboratory for the diagnosis of infectious Uveitis. The essential problem of the Uveitis is the etiological diagnosis since currently in 60% of cases no etiological diagnosis is brought out despite the deployment of routine diagnostic tests. The prognosis of the Uveitis is generally good but 15% approximately of Uveitis are evolving on a chronic mode which decreased faster than the Visual acuity of the eye reached that can lead to blindness in bilateral cases of Uveitis. Different works of the literature identified a few pathogenic microorganisms, viruses and bacteria as being responsible for uveitis, including within the particular framework of the endophtalmies. Recent work allowed to highlight the place of fastidious bacteria (Bartonella spp., Tropheryma whipplei, Rickettsia spp., Coxiella burnetii, Borrelia spp.) in these Uveitis. Despite all his investigations, is estimated that 20-30% of Uveitis likely to be of infectious origin are not documented by the methods used in routine. Our research project is to use a new microbiological diagnostic strategy of uveitis, allowing detection of the fastidious pathogens of infectious Uveitis who are not diagnosed by laboratory methods used in diagnostic routine. This new diagnostic strategy is to automatically detect the presence of a pathogen fastidious in cell culture using the same patient's serum to reveal a positive culture, based on the assumption that this serum contains antibodies specific pathogen tedious.

ELIGIBILITY:
Inclusion Criteria:

* Patient is more than 18 years old.

* Patient with a prescription of a microbiologic diagnostic of uveitis
* Patient who do not declined to have his medical records reviewed for research
* Patient with health insurance

Exclusion Criteria:

* Minor Patient ( age <18 years) (L. 1121-7 ) .

* Pregnant woman , parturient or nursing (L. 1121-5 ) .
* Patient major under guardianship (L. 1121-8 ) .
* Patient vital in emergency.
* Patient refusing to sign the informed consent form .
* Patient deprived of liberty under court order (L. 1121-6 ) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with an etiological diagnosis of Uveitis | 1 day

SECONDARY OUTCOMES:
Number of fastidious pathogenic germs detected | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance publique hôpitaux de marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided